CLINICAL TRIAL: NCT03736109
Title: Role of Copper-Albumin Complex in Treatment of Knee Osteoarthritis in Human:a Pilot Prospective Comparative Study
Brief Title: Role of Copper-Albumin Complex in Treatment of Knee Osteoarthritis in Human
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham I El-mahdy, Principal Investigator, Assiut University
Other Study IDs: Osteoarthritis
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Osteo Arthritis Knee
Keywords: Copper-Albumin Complex; Osteoarthritis; Syndecan 4; Substance P; hyaluronic acid; Insulin like growth factor; Nitric oxide
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I:: Thirty patients with knee osteoarthritis taking topical Copper-Albumin Complex cream
  Interventions: Genetic: Soluble and genetic biomarkers measurements
- Group II:: Thirty patients with knee osteoarthritis taking oral chondroprotective drugs
  Interventions: Genetic: Soluble and genetic biomarkers measurements

INTERVENTIONS:
Genetic: Soluble and genetic biomarkers measurements — Insulin-Like Growth Factor-1 and Coll2-1 gene expression will be measured by real time PCR. In addition, syndecan 4, hyaluronic acid, substance P and nitric oxide will be measured in plasma by ELISA

SUMMARY:
Osteoarthritis (OA) is one of the most common forms of degenerative joint disease and a major cause of pain and disability affecting the aging population. It is a significant burden in terms of cost as well as the health of society and individuals. Here in our study we will try to evaluate a novel therapeutic method by using topical copper-albumin complexes cream in treatment of osteoarthritis. Then all the biochemical changes will be measured beside the evaluation of topical copper-albumin complexes cream effectiveness in relieving symptoms of the OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a complex disease process involving the whole synovial joint. In OA articular cartilage is lost through a combination of degenerative and inflammatory phenomena, which are often accompanied by joint swelling, pain, stiffness and loss of joint mobility. The pathogenesis of OA is multifactorial and is considered to be a metabolically active process, predominantly due to the poor regenerative properties of articular cartilage after damage. The most commonly affected joint is the knee, and OA has a higher occurrence in older adults particularly women. Because patients generally present in the clinic after these symptoms of the illness develop, most treatment techniques for OA are designed to address these symptoms rather than cure the underlying disease. Current conservative treatments include lifestyle modification and pain medication (such as NSAIDs) which predominantly treat the illness (e.g., pain symptoms). There is also some promise in the use of chondroitin to decrease joint space narrowing in OA, thus treating the disease itself. Conversely, surgical intervention (partial or total joint replacement) is the preferred treatment method in end-stage disease leading to some relief of both the illness and disease.

Copper complexes can biochemically affect the cells and impinge upon metabolic pathways especially highly effective copper dependent enzymes, such as superoxide dismutase (SOD). It is predicted also that copper containing vitamins or biochemically active organic compounds such as amino acids and peptides or synthetic organic compounds in complexes can effectively scavenge superoxide radical. Additionally, recent studies showed that Cu (II) Bis (diethyldithiocarbamate) induced the expression of syndecan-4, a transmembrane heparan sulfate proteoglycan, in a dose- and time-dependent manner n via the activation of p38 mitogen-activated protein kinase. This submitted work has been designed to evaluate a copper chelating complex consisting of egg albumin and copper as one of the copper peptides that can be used as anti-inflammatory agent and chondroprotective in OA treatment that could be used as a substitute especially the currently used chondroprotective drugs are expensive and frequent using of drugs such as non-steroidal anti-inflammatory drugs (NSAIDs), known to be aggressive agents for gastric ulcer development.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes and over 40 years of age diagnosed with unilateral or bilateral symptomatic OA of the knee who met the criteria of the American College of Rheumatology (ACR).
* Patients who were rated grade II or III on the Kellgren and Lawrence (K&L) radiological scale [19].
* Patients with symptomatic OA with a global mean pain in the knee >40 mm on a Visual Analogue Scale (VAS) for pain assessment.

Exclusion Criteria:

* Women who were pregnant or breastfeeding
* Patients who were grade I or IV on K&L radiological scale.
* Patients who have had a prosthesis replaced in the 12 months prior to inclusion.
* Obesity

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Knee osteoarthritis patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-17 (Estimated); Primary Completion 2019-03-20 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
The mean difference of syndecan 4 expression and substance P before and after treatment | 2 months
  better understanding the efficacy of the Copper-Albumin Complex treatment for knee osteoarthritis

SECONDARY OUTCOMES:
Pain improvement | 2 months
  Visual Analog Score for pain

REFERENCES:
- [Background] Bai Z, Guo XH, Tang C, Yue ST, Shi L, Qiang B. Effects of Artesunate on the Expressions of Insulin-Like Growth Factor-1, Osteopontin and C-Telopeptides of Type II Collagen in a Rat Model of Osteoarthritis. Pharmacology. 2018;101(1-2):1-8. doi: 10.1159/000479160. Epub 2017 Sep 13. PMID 28898893
- [Background] Duncan C, White AR. Copper complexes as therapeutic agents. Metallomics. 2012 Feb;4(2):127-38. doi: 10.1039/c2mt00174h. Epub 2011 Dec 20. PMID 22187112
- [Background] Moller I, Gharbi M, Martinez Serrano H, Herrero Barbero M, Verges Milano J, Henrotin Y. Effect of chondroitin sulfate on soluble biomarkers of osteoarthritis: a method to analyze and interpret the results from an open-label trial in unilateral knee osteoarthritis patients. BMC Musculoskelet Disord. 2016 Oct 6;17(1):416. doi: 10.1186/s12891-016-1268-4. PMID 27716158
- [Background] Bay-Jensen AC, Thudium CS, Mobasheri A. Development and use of biochemical markers in osteoarthritis: current update. Curr Opin Rheumatol. 2018 Jan;30(1):121-128. doi: 10.1097/BOR.0000000000000467. PMID 29040157
- [Background] Ding H, Wu T. Insulin-Like Growth Factor Binding Proteins in Autoimmune Diseases. Front Endocrinol (Lausanne). 2018 Aug 30;9:499. doi: 10.3389/fendo.2018.00499. eCollection 2018. PMID 30214426